CLINICAL TRIAL: NCT02654405
Title: Sodium Butyrate As A Treatment For Improving Cognitive Function In Schizophrenia
Brief Title: Sodium Butyrate For Improving Cognitive Function In Schizophrenia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Nathan Kline Institute (NKI) decided not to accept study grant from Stanley Medical Research Foundation. because of budget considerations.
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Research Professor of Psychiatry, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 809383
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenic Disorders; Cognitive Function
Keywords: HDAC inhibitors; Inflammation
MeSH Terms: conditions — Schizophrenia; Inflammation | interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Butyrate (Experimental): 6.57 gms of sodium butyrate per day for 12 weeks
  Interventions: Dietary Supplement: Sodium Butyrate
- Placebo (Placebo Comparator): Placebo capsule with 2 mg of sodium butyrate for making taste or odor, (9 mg/day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium Butyrate — 6.57 gms of sodium butyrate per day for 12 weeks
  Arms: Sodium Butyrate
Other: Placebo — placebo capsules containing approximately 9 mg of sodium butyrate/day
  Arms: Placebo

SUMMARY:
The purpose of this grant is to evaluate the efficacy of sodium butyrate as a novel treatment for cognitive deficits in schizophrenia (SZ).

The proposal consists of a small preliminary open label study to assess tolerability and side effects of sodium butyrate in schizophrenic patients receiving antipsychotic treatment, followed by a larger double-blind study of the effects of sodium butyrate on cognitive function and symptoms in SZ patients who are not in an acute exacerbation of the primary symptoms and show continued cognitive deficits. Secondary aims will be to evaluate its effects on improving symptoms and functioning in SZ, and the relationship of the drug's clinical effects to epigenetic and inflammation related biochemical changes.

DETAILED DESCRIPTION:
The purpose of this grant is to evaluate the efficacy of sodium butyrate as a novel treatment for cognitive deficits in schizophrenia (SZ). Sodium butyrate is a short chain fatty acid and binds to the zinc site of histone deacetylases (HDAC). The inhibition of HDAC results in histone hyperacetylation.

The proposal consists of a small preliminary open label study to assess tolerability and side effects of sodium butyrate in schizophrenic patients receiving antipsychotic treatment ( in 5 patients with SZ treated with sodium butyrate for 8 weeks), followed by a larger double-blind study of the effects of sodium butyrate on cognitive function and symptoms, in SZ patients who are not in an acute exacerbation of the primary symptoms and show continued cognitive deficits. Secondary aims will be to evaluate its effects on improving symptoms and functioning in SZ, and the relationship of the drug's clinical effects to epigenetic and inflammation related biochemical changes. In the double-blind phase we plan a study at 3 sites: 2 US, 1 China, but only the US site at the Nathan Kline Institute ( NKI) will be active in the initial phase of the study.

We will provide a brief overview of the importance of these questions, some previous interventional treatment approaches, and the potential of HDAC inhibitors and sodium butyrate in particular to improve cognitive function.

The persistent cognitive deficits which can be appreciated across the course of SZ, from prodromal to chronic SZ, may be the most important underlying dysfunction in preventing functional, occupational, and social recovery in SZ compared to other symptom domains. There is no effective treatment for these cognitive deficits which persist after antipsychotic medication has reduced or resolved the positive symptoms of SZ. Although some exploratory studies of nicotinic agonist drugs showed promise for improvement of cognitive deficits associated with SZ , later larger and better-controlled studies with nicotinic agonist drugs have not shown markedly positive effects for this type of pharmacologic intervention, although one recent study is promising.

There is increasing interest in epigenetic mechanisms involving in DNA methylation and histone acetylation involved in the pathology underlying SZ and related disorders ). There is also interest in activation of inflammatory process as a part of the underlying pathophysiology of SZ, and there is research showing that effects on inflammatory markers may be partially mediated though epigenetic mechanisms of histone acetylation and DNA methylation. There is growing evidence that HDAC inhibitor drugs (HDACi) have properties of being cognitive enhancers and potential treatments for psychiatric disorders where cognitive deficits are prominent, such as SZ and Alzheimer's disease. Graff and Tsai suggest they may be particularly important in the process of promoting memory consolidation or conversion of short-term to longer- term memory and increasing memory retention or consolidation. Memory consolidation is demonstrated by the temporal gradient of retrograde amnesia (severity of amnesia most severe for events that occurred shortly before the amnesic event), as well as improvements in delayed recall of previously learned information after a retention interval. A specific deficit in memory consolidation has been demonstrated in SZ . Delayed recall performance may be used as an index of consolidation. For example, Goff et al found evidence of a beneficial effect of d-cycloserine on delayed but not immediate thematic recall using the Logical Memory Test (LMT) from the Revised Wechsler Memory Scale (WMS-R).

Sodium butyrate is a chemical compound found in foods and sold as a health food supplemental (a nutraceutical) which is a strong HDAC inhibitor (predominantly class I HDAC) and has anti-inflammatory and neuroprotective properties). Previous studies suggest it may have potential as a treatment for cognitive deficits in several psychiatric disorders, and have potential ameliorative effects on depression, and on human inflammatory diseases. Research with animal models show that sodium butyrate and phenylbutyrate have potential to improve cognition, including rescue of fear and spatial memories and enhancement of contextual memory, spatial memory and object recognition and improved memory in a mouse model of Alzheimer's disease. Sodium butyrate also decreased depressive-like behaviors in models of maternal deprivation and chronic stress . One human study with a butyrate congener improved cognitive outcome, including improvements in a test of working memory, in treatment of a urea cycle hyperammonia disorder. Sodium butyrate has also been used in clinical trials of inflammatory bowel diseases (Crohn's disease, ulcerative colitis) with positive effects on clinical state and also with improvement on indicators of inflammation . In the Crohn's disease study it also significantly decreased an immunological component interleukin-1 beta (IL-1 β). It has been used and sold widely as health food supplement nutraceutical in humans and has a good safety profile . It also reduces insulin resistance and lipid metabolic abnormalities as documented in both an animal model of fat induced insulin resistance and in an experimental human study preventing lipid induced insulin resistance . This effect may be relevant as a beneficial effect for metabolic abnormalities that are frequently reported in obese SZ. Sodium butyrate is lipophilic compound that passes the blood-brain barrier. This is reported in previous studies and reviews stating that sodium butyrate crosses the blood brain barrier). For example, in a mouse model oral sodium butyrate increased histone acetylation both in brain and periphery. This fulfills a criterion the Stanley granting organization requests be reported for proposed pharmacological studies.

The above background provides a rationale for a trial of sodium butyrate as a cognitive enhancer in SZ.

The specific aims of the double-blind will be to test the following hypotheses.

Primary Aim:

1. Treatment with sodium butyrate will improve cognition in SZ as measured by the composite and domain scores of the Measurement and Treatment Research to Improve Cognition in Schizophrenia battery (MATRICS [MCCB]) . The primary outcome measure will be the MCCB composite score.

   Secondary Aims:
2. Treatment with sodium butyrate will improve memory consolidation as measured by delayed recall performance.
3. Improvement in cognitive function induced by sodium butyrate in SZ will be correlated with improvement in a measure of performance on real world functional tasks as assessed by the University of California San Diego (USCD) Performance- Based Skills Assessment Battery (UPSA).

We will also explore whether improvement in cognition is related to change in HDAC activity in peripheral blood cells and changes in inflammatory makers in the blood (CRP, IL-1 β ), and assess whether there is any improvement in psychopathology as measured by PANSS scale.

The study will be conducted in two phases, an open-label study of the safety and tolerability of sodium butyrate in patients with schizophrenia followed by a randomized placebo controlled experimental study of the effects of adjunctive 6.57 gms of sodium butyrate per day for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis by DSM-5 (Diagnostic Statistical Manual) diagnosis of SZ or schizoaffective disorder (SA), by consensus diagnosis using chart histories and interviews.
2. Age 18-60 years of age.
3. Patients will be stably treated with antipsychotic medications and are not in acute illness exacerbation of their symptoms.

   For the double-blind phase only qualification for cognitive deficits will use the following criteria:
4. Subjects will have baseline MCCB battery scores which meet the following criteria. Subjects will meet the following cognitive performance criteria: a). Maximum performance level: Performance at least 1.0 standard deviation (SD) from perfect on the following three measures: Letter-number span (< 24), Hopkins Verbal Learning Test (HVLT) total (<31), Continuous Performance Test (CPT) d-prime (< 3.47) and b.
5. Minimum performance level: subject must be able to validly complete the baseline MATRICS assessment.

Exclusion Criteria:

1. History of mental retardation or pervasive developmental disorder.
2. Subjects with a current serious neurological/central nervous system (CNS) disorder (such as seizure disorder, stroke or multiple sclerosis) or brain trauma.
3. Current treatment with valproic acid, butyrate drugs, sulforaphane, or other drugs or chemicals known to have high HDAC inhibitory activity.
4. Pregnancy.
5. Severe unstable current medical condition.
6. Current suicidal or homicidal thoughts.
7. Current alcohol or substance abuse (other than nicotine or occasional marijuana) in the last month.
8. Subjects with diagnosis of congestive heart failure, or those on sodium restricted diet.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in MATRICS Battery Score | Baseline, week 6, up to 12 weeks
  MATRICS Cognitive Battery

SECONDARY OUTCOMES:
Change from baseline Logical Memory test score | baseline, 12 weeks
  Logical Memory Test for longer Term Memory
Change from baseline in PANSS Total Score | baseline, 6 weeks, up to 12 weeks
  PANSS symptom rating scale
Change from baseline in PASAT Score | baseline,6 weeks, up to 12 weeks
  Alternate working memory test
change from baseline in UPSA Total score | baseline, 12 weeks
  USCD (University of California San Diego) Performance- Based Skills Assessment Battery

OTHER OUTCOMES:
Change from baseline in Side-Effect Scale Score | baseline,2 weeks, 6 weeks, up to 12 weeks
  Patient self-report of side-effects of active or placebo medication
Change from baseline in clinical laboratory measures | baseline, 12 weeks
  common clinical laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, M.D., Ph.D, Principal Investigator — Nathan Kline Institute for Pstychiatric Research
Locations (1):
- Nathan Kline Insitute for Psychiatric Research, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Stanley foundation requests: Based on the terms of your award, Stanley Medical Research Institute (SMRI) now requires submission of the individual patient data from all SMRI funded studies. In order to make the process as efficient as possible and provide a secure location for study data, National Institute of Mental Health (NIMH) is graciously allowing SMRI access to their National Database for Clinical Trials (NDCT) to collect and house data